CLINICAL TRIAL: NCT00321425
Title: Ultrasound Guidance Vs. Electrical Nerve Stimulation for Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rikshospitalet University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: S-05240
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2007-10

CONDITIONS: Hand Surgery; Brachial Plexus Block
MeSH Terms: interventions — Brachial Plexus Block; Transcutaneous Electric Nerve Stimulation

INTERVENTIONS:
Procedure: brachial plexus block
Procedure: ultrasound guidance
Procedure: electrical nerve stimulation

SUMMARY:
In an observer-blinded study ultrasound guidance and electrical nerve stimulation will be compared for lateral sagital infraclavicular blocks (LSIB). Block effectiveness, time consumption and patient acceptance will be registered in 80 patients. Ultrasound guidance may cause less discomfort and could be less time consuming than electrical nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Infraclavicular brachial plexus block
* Hand surgery

Exclusion Criteria:

* ASA > 2
* Block assessment impossible
* Allergy to local anesthetic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-05

PRIMARY OUTCOMES:
Block effectiveness, time consumption; patient acceptance, discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Axel R Sauter, MD, Principal Investigator — Department of Anaesthesiology, Rikshospitalet University Hospital; Øivind Klaastad, MD, Principal Investigator — Department of Anaesthesiology, Rikshospitalet University Hospital; Audun Stubhaug, MD, Study Chair — Department of Anaesthesiology, Rikshospitalet University Hospital
Locations (1):
- Department of Anaesthesiology, Rikshospitalet University Hospital, Oslo, Oslo County, Norway